CLINICAL TRIAL: NCT07377838
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of ADSTEM Inj. for Moderate to Severe Subacute and Chronic Atopic Dermatitis Patients
Brief Title: Study of ADSTEM Injection for Patients With Moderate to Severe Subacute and Chronic Atopic Dermatitis
Acronym: ADSTEM Inj
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: EHL Bio Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AD-CP-23-1
Record Dates: First submitted 2026-01-22; First posted 2026-01-30 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Atopic Dermatitis
Keywords: Adipose Derived Mesenchymal Stem cell; AD; Inflammatory disease; ADMSC; Stem cell; ehlbio
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADSTEM Inj. (Experimental)
  Interventions: Biological: ADSTEM Inj.
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: ADSTEM Inj. — hAD-MSC 1.0x10^8 cells
  Arms: ADSTEM Inj.
Drug: Placebo — 0.9% Normal Saline Inj.
  Arms: Placebo

SUMMARY:
Study of ADSTEM Injection for Patients with Moderate to Severe Subacute and Chronic Atopic Dermatitis

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 19 to 70 years at the time of informed consent.
2. Diagnosis of atopic dermatitis according to the Hanifin and Rajka criteria at screening.
3. History of atopic dermatitis for at least 24 weeks prior to screening.
4. Moderate-to-severe atopic dermatitis at screening, defined as:

   * EASI score ≥16
   * SCORAD score ≥25
   * Body Surface Area (BSA) involvement ≥10%
   * vIGA score ≥3
5. Inadequate response to prior standard topical and/or systemic treatments for atopic dermatitis, or inability to receive such treatments due to safety concerns.
6. Voluntary written informed consent provided.

Exclusion Criteria:

1. Presence of clinically significant comorbidities at screening, including:

   * Active infection requiring antimicrobial treatment within 2 weeks prior to baseline, or superficial skin infection within 1 week prior to baseline;
   * Skin diseases that require ongoing treatment or may interfere with safety or efficacy assessments;
   * Uncontrolled asthma requiring oral corticosteroids;
   * Positive test results for hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV), or syphilis;
   * Other uncontrolled or clinically significant medical conditions that may affect study participation or assessments;
   * Clinically significant abnormal laboratory results at screening (e.g., AST or ALT > 3 × ULN, serum creatinine > 2 × ULN).
2. History of prohibited treatments prior to baseline, including:

   * Use of JAK inhibitors within 4 weeks;
   * Use of biologic therapies for atopic dermatitis within 12 weeks;
   * Use of systemic immunosuppressants, immunomodulators, or systemic corticosteroids within 4 weeks;
   * Use of topical corticosteroids, topical PDE-4 inhibitors, or topical calcineurin inhibitors within 2 weeks;
   * Participation in another clinical trial with an investigational drug or device within 4 weeks prior to screening;
   * Prior treatment with cell therapy or gene therapy.
3. History of malignancy within 5 years prior to screening, except adequately treated non-melanoma skin cancer without recurrence.
4. History of tanning within 4 weeks prior to baseline.
5. Pregnant or breastfeeding women, or women planning pregnancy during the study period.
6. Women of childbearing potential who are unwilling to use adequate contraception from the time of informed consent through the end of the study.
7. Known or suspected hypersensitivity to the investigational product or any of its components.
8. Any other condition that, in the investigator's judgment, makes the participant unsuitable for participation in the study.

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2026-06 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants who achieve a score of 0 or 1 on the validated Investigator's Global Assessment (vIGA) scale at Visit 6, and demonstrate at least a 2-point reduction from baseline(Visit 2) | From baseline to Weeks 16
  validated Investigator's Global Assessment [vIGA], 0-4, higher scores indicate worse disease severity

SECONDARY OUTCOMES:
Change from baseline (Visit 2) in vIGA score | From baseline to Weeks 4, 8, 12, 16, 20, and 24
Percentage of participants with a vIGA score reduction of 1 point or ≥2 points from baseline (Visit 2) | From baseline to Weeks 4, 8, 12, 16, 20, and 24
Percentage of participants with a vIGA score of 0 or 1 at Week 24 | From baseline to Week 24
Percentage of participants with a ≥50% reduction in total EASI score from baseline (Visit 2) | From baseline to Weeks 4, 8, 12, 16, 20, and 24
  Eczema Area and Severity Index [EASI], 0-72, higher scores indicate worse disease severity
Percentage of participants with a ≥75% reduction in total EASI score from baseline (Visit 2) | From baseline to Weeks 4, 8, 12, 16, 20, and 24
Percentage of participants with a ≥90% reduction in total EASI score from baseline (Visit 2) | From baseline to Weeks 4, 8, 12, 16, 20, and 24
Change from baseline (Visit 2) in total EASI score | From baseline to Weeks 4, 8, 12, 16, 20, and 24
Percentage of participants with a ≥50% reduction in total SCORAD score from baseline (Visit 2) | From baseline to Weeks 4, 8, 12, 16, 20, and 24
  Scoring Atopic Dermatitis [SCORAD], 0-103, higher scores indicate worse disease severity
Percentage of participants with a ≥75% reduction in total SCORAD score from baseline (Visit 2) | From baseline to Weeks 4, 8, 12, 16, 20, and 24
Change from baseline (Visit 2) in total SCORAD score | From baseline to Weeks 4, 8, 12, 16, 20, and 24
Change from baseline (Visit 2) in individual SCORAD item scores | From baseline to Weeks 4, 8, 12, 16, 20, and 24
Change from baseline (Visit 2) in DLQI score | From baseline to Weeks 8, 16, and 24
  Dermatology Life Quality Index [DLQI], 0-30, higher scores indicate worse quality of life
Percentage of participants using rescue medication, number of uses, and total amount used | From Week -6 (Visit 1) to Weeks 4, 8, 12, 16, 20, and 24

IPD SHARING:
Plan to Share IPD: No